CLINICAL TRIAL: NCT00382239
Title: A Dose Response Study to Assess the Effect on Glucose Control and Safety and Tolerability of LY2148568 in Japanese Patients With Type 2 Diabetes Who Are Treated With Oral Antidiabetic(s) But Not Well Controlled
Brief Title: A Study to Assess the Effect on Glucose Control and Safety and Tolerability of LY2148568 In Japanese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-JE-GWAV
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; LY2148568; Lilly; Amylin; Japan
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exenatide 5 mcg/exenatide 10 mcg (Experimental)
  Interventions: Drug: exenatide (LY2148568)
- Exenatide 5 mcg/exenatide 5 mcg (Experimental)
  Interventions: Drug: exenatide (LY2148568)
- Exenatide 2.5 mcg/exenatide 2.5 mcg (Experimental)
  Interventions: Drug: exenatide (LY2148568)
- Placebo/placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: exenatide (LY2148568) — subcutaneous injection twice daily, 5 mcg for 4 weeks, then 10 mcg for 8 weeks
  Other Names: Byetta
  Arms: Exenatide 5 mcg/exenatide 10 mcg
Drug: exenatide (LY2148568) — subcutaneous injection twice daily, 5 mcg for 4 weeks, then 5 mcg for 8 weeks
  Other Names: Byetta
  Arms: Exenatide 5 mcg/exenatide 5 mcg
Drug: exenatide (LY2148568) — subcutaneous injection twice daily, 2.5 mcg for 4 weeks, then 2.5 mcg for 8 weeks
  Other Names: Byetta
  Arms: Exenatide 2.5 mcg/exenatide 2.5 mcg
Drug: Placebo — subcutaneous injection twice daily, 0.02 mL to 0.04 mL
  Arms: Placebo/placebo

SUMMARY:
This study will examine the response of several doses of LY2148568 (exenatide) and assess the effect on glucose control and safety and tolerability in Japanese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes.
* Have a body weight of >=50 kg.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have participated in this study previously, or any other study using exenatide or other GLP-1 analogs.
* Are treated with any exogenous insulin within 3 months of screening.
* Are continuously treated with any of the following excluded medications within 3 months of screening (more than 7 days per 1 month): *drugs that directly affect gastrointestinal motility, including Nauzelin® (domperidone), Primperan®/Terperan® (metoclopramide), Ganaton® (itopride), Acenalin® (cisapride), Gasmotin® (mosapride), or Cerekinon® (trimebutine).
* Have characteristics contraindicating for concomitant medication, according to product-specific label.
* Have severe allergy or hypersensitivity to any drug.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Week 12 | Baseline, Week 12
  Assess dose response effect on glucose control as measured by HbA1c among four doses (2.5 μg, 5 μg, 10 μg, and placebo) of subcutaneous injection of exenatide, twice daily before meals in the morning and evening, for 12 weeks

SECONDARY OUTCOMES:
Proportion of subjects achieving HbA1c <7% at Week 12 | 12 weeks
  Total number of subjects achieving HbA1c <7% at Week 12
Changes in fasting blood glucose from Visits 3 to 7 | Baseline, Week 12
  Changes in fasting blood glucose from Baseline (Visit 3) to Week 12 (Visit 7)
Change in Serum lipids from Baseline to Week 12 | Baseline, Week 12
  Changes in serum lipids (total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides) from Baseline (Visit 3) to Week 12 (Visit 7)
Changes in body weight, waist size and waist/hip ratio from Baseline to Week 12 | Baseline, Week 12
  Changes in body weight, waist size and waist/hip ratio from Baseline (Visit 3) to Week 12 (Visit 7)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (14):
- Japan (14):
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kanagawa
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Nagano
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Tokyo

REFERENCES:
- [Result] Kadowaki T, Namba M, Yamamura A, Sowa H, Wolka AM, Brodows RG. Exenatide exhibits dose-dependent effects on glycemic control over 12 weeks in Japanese patients with suboptimally controlled type 2 diabetes. Endocr J. 2009;56(3):415-24. doi: 10.1507/endocrj.k08e-296. Epub 2009 Feb 4. PMID 19194050
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356